CLINICAL TRIAL: NCT02731456
Title: Effect of High Altitude Exposure, Acclimatization and Re-exposure on Psychomotor Performance and Sleep Quality in Lowlanders
Brief Title: Effect of High Altitude Exposure, Acclimatization and Re-exposure on Psychomotor Performance in Lowlanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Poulin (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Marc Poulin, Professor, University of Calgary
Organization: University of Calgary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB15 - 2709_MOD1
Record Dates: First submitted 2016-04-03; First posted 2016-04-07 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Effect of High Altitude
Keywords: high altitude; cognition; sleep
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altitude exposure (Experimental): Acute high altitude exposure followed by 8 day acclimatization and re-exposure for 8 days after 6 days at low altitude.
  Interventions: Other: altitude exposure

INTERVENTIONS:
Other: altitude exposure — altitude exposure

SUMMARY:
Prospective interventional trial in lowlanders evaluating the effect of acute exposure, acclimatization and re-exposure to high altitude on psychomotor vigilance to measure sustained attention.

DETAILED DESCRIPTION:
Baseline measurements will be performed in Santiago de Chile, 520 m, over the course of 3 days. Participants will then travel by commercial airline (2 h flight) and by bus (2 h ride) to the ALMA base camp located at 2900 m near San Pedro de Atacama, northern Chile. Participants will stay there for the next 7 nights and they will spend the days (6 total; 6-8 h daily) at the telescope station at 5050 m while undergoing testing as described above at the first and the last day at 5050m. Daily transports from 2900 to 5050 m will be by car (1 h ride, one way). After the first 7 day altitude sojourn participants will return to the Santiago area (520 m) for a 7 day recovery period. A second altitude sojourn with an identical schedule as the one described above and a final low altitude stay of 3 days will follow.

ELIGIBILITY:
Inclusion Criteria:

* born, raised and currently living <1300m
* No overnight stays at altitudes >1500m 4 weeks before the study

Exclusion Criteria:

* previous altitude intolerance <3000m
* pregnancy
* health impairment, which requires regular treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Sustained attention measured by a visual pychomotor vigilance test (PVT) | Low altitude dojourn at 520m; forst sojourn at 5050m Day 2, 7; second sojourn at 5050m Day 2, 7
  Change in psychomotor response speed across two cycles of altitude exposure, comparing 5050m to 520m.

SECONDARY OUTCOMES:
Indices of sleep quality measured by actigraphy (total sleep time, sleep efficiency, sleep latency | Low altitude dojourn at 520m; forst sojourn at 5050m Day 2, 7; second sojourn at 5050m Day 2, 7

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Poulin, PhD, DPhil, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No